CLINICAL TRIAL: NCT01858376
Title: Effect Of Capros Supplementation On Cardiovascular Disease Risk Factors In Humans
Acronym: Capros
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chandan K Sen (Other)
Collaborators: Natreon, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chandan K Sen, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012H0381
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Results first posted 2015-11-09 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2017-10

CONDITIONS: Hyperlipidemia
Keywords: LDL cholesterol; anti-hyperlipidemic; hyperlipidemic; Capros; Natural Supplement
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capros dietary supplement (Other): Subjects will take Capros supplement (1 capsule) twice a day for 12 weeks.The subjects then will have blood drawn seven times throughout the course of the study.
  Interventions: Dietary Supplement: Capros dietary supplement

INTERVENTIONS:
Dietary Supplement: Capros dietary supplement — Study participants will have 2 to 3 baseline blood draws, 3 blood draws while taking Capros supplements and 2 wash out blood draws after finishing 12 weeks of Capros supplementation. Participants will attend 7 to 8 study visits (depending on number of baseline visits needed) and at each visit participants will have their blood drawn as well as height, weight, blood pressure, and pulse measured.

SUMMARY:
The hypothesis of this study is that the natural supplement Capros will decrease LDL levels, platelet aggregation, and serum concentrations of high sensitivity C-reactive protein in humans at risk for cardiovascular disease.

DETAILED DESCRIPTION:
A non-randomized, longitudinal study to determine the effect of Capros supplementation on a lipid profile, platelet aggregation and high-sensitivity C - reactive protein in 30 volunteers at risk for cardiovascular disease.

-Herbal Polyphenols/Antioxidants: Role in Cardiovascular Disease Prevention: Phenolic compounds are dietary antioxidants found in plants that are shown to inhibit LDL oxidation, inhibit platelet aggregation and adhesion, decrease total and LDL cholesterol, and induce endothelium-dependent vaso-relaxation. [Lapointe, Vita, and Mendes]. Epidemiologic studies suggest that higher polyphenol intake from fruits and vegetables is associated with decreased risk for cardiovascular disease. Among the numerous plausible mechanisms by which polyphenols may offer cardiovascular protection, improvement of the endothelial function and inhibition of angiogenesis and cell migration and proliferation in blood vessels have been the focuses of recent studies. Antioxidants in polyphenols, in addition to protecting LDL cholesterol against oxidation, may act at a vascular cell level by limiting cellular production of reactive oxygen species, and, thus, cell-mediated LDL oxidation. In traditional Indian medicine, the gooseberry (Phyllanthus emblica) has been used for thousands of years as an effective source of polyphenols and antioxidants. "P. emblica is considered beneficial against various diseases namely cancer, diabetes, liver treatment, and various other diseases."[Hiraganahalli]. Capros®, from Natreon, Inc., is a cascading antioxidant ingredient derived from Phyllanthus emblica. It has been used in cosmetics and food-and-beverage formulations in many countries, and, based on extensive scientific research, also shows particular promise as a dietary supplement.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21-70 years of age
* BMI 25-35

Exclusion Criteria:

* BMI > 35 OR < 25
* Smokers
* Individuals who are deemed unable to understand the procedures, risks and benefits of the study, i.e. Informed consent will be excluded
* Females who are pregnant as well as individuals who are therapeutically immuno-compromised will also be excluded in order to minimize the risk to such individuals (and fetus) and to decrease statistical variability and to minimize potential of confounders.
* Candidates for inclusion into the study will not include individuals as defined in 45 CFR 46 Subparts B, C and D, nor from any other population which may be considered vulnerable. Pregnant women are excluded to minimize the risk to such individuals (and fetus) and to decrease statistical variability and to minimize potential of confounders.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Brieger K, Schiavone S, Miller FJ Jr, Krause KH. Reactive oxygen species: from health to disease. Swiss Med Wkly. 2012 Aug 17;142:w13659. doi: 10.4414/smw.2012.13659. eCollection 2012. PMID 22903797
- [Result] Rigaud JL, Gulik-Krzywicki T, Seigneuret M. Freeze-fracture electron microscopy study of bacteriorhodopsin oligomerization. Prog Clin Biol Res. 1988;273:99-104. No abstract available. PMID 3420138
- [Result] Carchietti E, Baldassarre M, Penco T, Leonardi M. Iopamidol 300-induced epilepsy: intensive treatment and pathogenic hypothesis. Neuroradiology. 1988;30(3):256-7. doi: 10.1007/BF00341838. PMID 3405414
- [Result] Taleb A, Tsimikas S. Lipoprotein oxidation biomarkers for cardiovascular risk: what does the future hold? Expert Rev Cardiovasc Ther. 2012 Apr;10(4):399-402. doi: 10.1586/erc.12.32. No abstract available. PMID 22458571
- [Result] Stoclet JC, Chataigneau T, Ndiaye M, Oak MH, El Bedoui J, Chataigneau M, Schini-Kerth VB. Vascular protection by dietary polyphenols. Eur J Pharmacol. 2004 Oct 1;500(1-3):299-313. doi: 10.1016/j.ejphar.2004.07.034. PMID 15464042
- [Result] Gokce N, Frei B. Basic research in antioxidant inhibition of steps in atherogenesis. J Cardiovasc Risk. 1996 Aug;3(4):352-7. doi: 10.1177/174182679600300403. PMID 8946264
- [Result] Hiraganahalli BD, Chinampudur VC, Dethe S, Mundkinajeddu D, Pandre MK, Balachandran J, Agarwal A. Hepatoprotective and antioxidant activity of standardized herbal extracts. Pharmacogn Mag. 2012 Apr;8(30):116-23. doi: 10.4103/0973-1296.96553. PMID 22701284
- [Result] Brauer K, Schober W, Winkelmann E, Garey LJ. Topographic differences in retinal axons in the dorsal lateral geniculate nucleus of the rat: a quantitative reexamination using anterograde transport of horseradish peroxidase. Exp Brain Res. 1988;69(3):481-8. doi: 10.1007/BF00247302. PMID 3371432
- [Derived] Khanna S, Das A, Spieldenner J, Rink C, Roy S. Supplementation of a standardized extract from Phyllanthus emblica improves cardiovascular risk factors and platelet aggregation in overweight/class-1 obese adults. J Med Food. 2015 Apr;18(4):415-20. doi: 10.1089/jmf.2014.0178. Epub 2015 Mar 10. PMID 25756303

RESULTS

PARTICIPANT FLOW:
Groups:
- Capros Dietary Supplement: Subjects will take Capros supplement (1 capsule) twice a day for 12 weeks.The subjects then will have blood drawn seven times throughout the course of the study.
  Capros dietary supplement: Study participants will have 2 to 3 baseline blood draws (as needed), 3 blood draws while taking Capros supplements and 2 wash out blood draws after finishing 12 weeks of Capros supplementation. Participants will attend 7 to 8 study visits (depending on number of baseline visits needed) and at each visit participants will have their blood drawn as well as height, weight, blood pressure, and pulse measured.
Period: Overall Study
Arm/Group | Capros Dietary Supplement
Started | 24
Completed | 20
Not Completed | 4
Not completed — Dropped d/t lab work not fitting criter | 4

BASELINE CHARACTERISTICS:
Arm/Group | Capros Dietary Supplement
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 28.57 (2.71)
Blood Pressure Systolic [Mean (Standard Deviation); unit: mm Hg] | 116.87 (7.19)
Height [Mean (Standard Deviation); unit: cm] | 171 (9.38)
Weight [Mean (Standard Deviation); unit: lbs.] | 185.19 (27.67)
Blood Pressure Diastolic [Mean (Standard Deviation); unit: mm Hg] | 76.91 (6.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lipid Profile
Description: Blood lipid panel including HDL, LDL, total cholesterol. Looking at Baseline to 12 weeks on supplement with a two week washout period
Time Frame: Baseline and 14 weeks
Population: number of participants analyzed is different from the participant flow module due to subjects who self reported non-compliance from pill count of the supplements and their data was not able to be used for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Capros Dietary Supplement
Number analyzed (Participants) | 9
mg/dl
  HDL cholesterol | 4.20 [-6.21 to 14.62]
  LDL cholesterol | 3.37 [-7.62 to 14.36]
  Total Cholesterol | -0.06 [-0.34 to 0.22]

2. Secondary Outcome: Changes in High-Sensitivity C-reactive Protein
Description: High-Sensitivity C-reactive Protein analysis in blood. Looking at Baseline to 12 weeks on supplement with a two week washout period
Time Frame: Baseline and 14 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Capros Dietary Supplement
Number analyzed (Participants) | 15
mg/dl | 0.07 [-0.44 to 0.58]

3. Secondary Outcome: C-reactive Protein
Description: C-reactive protein in blood as measured in a standard hospital laboratory. 12 weeks on supplementation data presented.
Time Frame: Baseline and 14 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Capros Dietary Supplement
Number analyzed (Participants) | 15
mg/L | 1.61 (1.18)

4. Secondary Outcome: Changes From Baseline in Platelet Aggregometry
Description: Adenosine Diphosphate (ADP), Arachidonic acid (AA), and Collagen (unsure about the specific type of collagen) agonists will be measured using optical platelet aggregometry. Looking at Baseline to 12 weeks on supplement with a two week washout period
Time Frame: Baseline and 14 weeks
Measure: Mean (95% Confidence Interval); unit: maximum % aggregation
Arm/Group | Capros Dietary Supplement
Number analyzed (Participants) | 12
maximum % aggregation
  ADP | 3.34 [-12.56 to 19.23]
  AA | -9.56 [-32.15 to 13.03]
  Collagen | 15.76 [-6.86 to 38.37]

ADVERSE EVENTS:
Time Frame: 14 weeks from baseline of beginning the supplement to 12 weeks of ending supplementation, followed by 2 weeks of washout.
Arm/Group | Capros Dietary Supplement
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No